CLINICAL TRIAL: NCT02274948
Title: Effects of Metformin on Body Weight, Composition and Metabolic Derangements in Obese Children. A Randomized Clinical Trial
Brief Title: Use of Metformin in Treatment of Childhood Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colombo (Other)
Responsible Party: Principal Investigator, Pujitha Wickramasinghe, Professor in Paediatrics, University of Colombo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC-13-143
Record Dates: First submitted 2014-10-19; First posted 2014-10-27 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): 8-10.99 year old children received metformin. Initially children given 250mg of metformin daily for a week and increased to 250mg twice daily for a week and then to 500 mg twice daily there after. 11-16 year old children received 500mg of metformin daily initially for one week which increased to 500mg twice daily for a week and then to 1g twice daily. The medication was continued for 12 months.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): A placebo tablet which is physically similar to metformin tablets will be given in a similar manner as described above.
  Metformin and placebo is manufactured by the State Pharmaceutical Manufacturing Corporation (SPMC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin in the form of 500mg tablets were administer to the Metformin group
  Other Names: Generic Metformin Produced by SPMC, Sri Lanka
  Arms: Metformin
Drug: Placebo — A Placebo tablet physically and chemically similar to Metformin tablets except for the absence of the active ingredient was used
  Other Names: Placebo manufactured by SPMC, Sri Lanka
  Arms: Placebo

SUMMARY:
This study expects to evaluate the use of metformin in the management of obese children. Insulin resistance among obese Sri Lankan children (south Asian origin) is high, which had been shown in the investigators previous work.

This study will look at the effect of metformin on changes in insulin resistance, fatty liver state, body fat content, BMI and other metabolic derangement.

DETAILED DESCRIPTION:
1. General objective To study the prevalence of Non Communicable Disease (NCD) related metabolic derangements among obese children and assess the outcome of two different management (metformin vs placebo alongside dietary and physical activity changes) modalities among 8 to16 year old obese children living in Negombo educational division of Negambo educational zone of Gampaha district in Sri Lanka.

1.1 Specific objectives

1. To study the prevalence of obesity related metabolic derangements among obese children.
2. To compare the effectiveness of the use of metformin vs placebo in the change of fat content and BMI among obese children.
3. To compare the effectiveness in the use of metformin vs placebo in the reversal of insulin resistance and metabolic derangements among obese children.

2 Methods 2.1 Study design A double blind randomized prospective placebo control study

2.2 Subjects and Study setting Obese (more than +2 Standard Deviation (SD) of BMI to age on World Health Organization (WHO) standards) school children from Negombo educational zone of district of Gampaha.

Obese children had been identified in a separate screening programme (it will be carried out during Sep-Dec 2013 and Sri Lanka College of Paediatricians, ethical review committee has approved the study protocol) carried out in this same educational division and are invited to participate in this study. Children not of Sri Lankan origin or who are not planning to live in Sri Lanka during the next one year or has a secondary underlying cause for the overweight/obesity, will be excluded.

Parents will be informed about the importance of participating in the study from the point of receiving treatment as well as participating in the research (written information sheet will given) and informed written consent from parents/guardians and assent from child will be obtained. Any parent, child who wishes not to participate will allowed doing so.

2.3 Sample size and sampling method: All children who were detected to be obese in a previous screening programme will be invited and a minimum sample size of 120 children will be recruited.

The sample size is calculated, that among obese children, a total sample size of 60 participants would detect a between-group difference of 0.09 BMI SD score units (approximately equivalent to a 2 kg/m2 difference) with 80% power. Participant accrual was set at 120 participants to allow as much as 50 percent loss to follow-up. However, the investigators will take maximum effort to trace the patients.

2.4 Measurements: These children will be invited to participate in a follow up programme as part of clinical service as well as research. Their parents will be informed to bring their children to the Loins Club of Negambo Host, Diabetes Screening and Vocational Training Centre, Negambo by appointment.

Measurements will be done at the Loins Club of Negambo Host, Diabetes Screening and Vocational Training Centre, Negamboafter an overnight fast. Height, weight, waist circumference and hip circumference will be measured. Percentage fat mass will be measured using Bio Electrical Impedance (BIA) assay using platform type InBody 230 instrument (InBody®, Biospace, South Korea). Once the impedance value is measured, total body water will be calculated using the locally validated BIA prediction equation (Wickramasinghe et al 2008). From Total Body Water (TBW), Fat Free Mass (FFM) and hence Fat Mass (FM) was calculated using age and gender specific water content of FFM (Lohman, 1989). Blood pressure will be measured using a mercury sphygmomanometer in seated position after 10-15 minute rest. Male and female children will be assessed by trained male and female investigators respectively.

Metabolic derangements will be assessed by means of: total cholesterol, LDL-C levels, HDL-C levels, triglyceride, insulin, Alanine amino transferase (ALT) and Aspartate amino transferase (AST) (8ml of blood into a plain bottle) fasting blood sugar (2ml of blood into a NaF containing bottle). Oral Glucose Toerance Test (OGTT) test will be done after giving anhydrous glucose 1.75g (1.92g of monohydrous glucose) to max of 75g (max 82.5g of monohydrous glucose) and blood will be taken 2 hour later for random blood sugar (2ml of blood into a NaF containing bottle) and serum insulin (2ml of blood into a plain bottle). Serum will be separated immediately and stored at -20 degree of Celcius and analysis will be done at Loins Club of Negambo Host, Diabetes Screening and Vocational Training Centre, Negambo in batches. Blood will be drawn after applying lignocaine (Emla®) anesthetic cream.

Insulin resistance will be calculated using Homeostatic model Insulin Resistance (HOMA-IR= fasting blood sugar × fasting insulin ÷ 22.5) (Matthews et al 1985). An Ultra sound scan of abdomen will be done to identify hepatic steatosis by a consultant radiologist.

Pubertal staging will be assessed using visual charts (Morris and Udry 1980). Girls will be shown a diagram depicting different stages of growth of breasts and pubic hair and ask them to match it with their own (whenever necessary will seek mother's assistance). Similarly boys are shown diagrams of external genitalia and pubic hair and to match with their own. The size of the testis will be measure by the examiner using Prader orchidometer. If both subject and parents were not sure of the staging, with consent, the examiner would examine and the correct pubertal stage assessment would be made. Measurements and examinations in girls and boys will be carried out by female and male investigators respectively.

The whole project will be closely supervised by a two Consultant paediatricians and after the completion of study children who need follow up will be provided the services or if they wish to be followed up at a different institute, would be referred with a complete report.

2.5 Randomization: Once obesity and overweight is diagnosed and investigated, they will be randomly assigned to either of one management protocol on a 1:1 basis. Children will be categorized according to gender and age groups; 8-10.99; 11-13.99; 14-16 years. Using a grid for each age of each sex, sequentially they will be allocated to receive management protocol I or II. Only the field investigators will have information to the allocation. That is; Group I Structured diet + Physical activity+ Metformin Group II Structured diet + Physical activity + Placebo

Dietary advice will be given by a trained nutritionist. It will be based on food based dietary guidelines produced by Ministry of Health (Jayatissa and Wickramasinghe, 2011). Age based portion size guide will be given to parents and children and guide them on the volume they should be eating.

Physical activity training will be conducted by a qualified physical activity instructor. A daily physical activity routine of 20-30 minutes will be given to each student. The programme would be of 3 different types based on their age (11-13 and 14-16. The workout programme will be changed every month in order to break the monotony. There will 4 such different workout schedules.

Medication: 8-10.99 year old children will receive metformin. Initially children will be given 250mg of metformin daily for a week and increased to 250mg twice daily for a week and then to 500 mg twice daily there after. 11-16 year old children will receive 500mg of metformin daily initially for one week which will be increased to 500mg twice daily for a week and then to 1g twice daily. Children will be asked to take medication with their morning and evening meals to reduce gastro intestinal side effects and risk of hypoglycaemia. Response to medication will be evaluated before each dose revision and will monitor for all possible adverse events.

The study will be monitored by a Data and Safety Monitoring Committee comprising of a Paediatrician, Paediatric Endocrinologist and a Bio- Statistician.

Both the nutritionist and physical trainer will be blinded to the medication children will be receiving.

A control group with no treatment will not be employed as it will be unethical not to do any intervention when the diagnosis of obesity is made. A placebo is given to overcome any psychological effects of giving medication. metformin and Placebo will be manufactured by the State Pharmaceutical Manufacturing Company (SPMC). The placebo tablet will be similar to metformin in all aspects except for containing the active pharmacological compound.

These children will be reviewed two weeks after commencement of therapy and dose will be revised and thereafter monthly in order to ensure compliance and identify any adverse events and address issues. In additionally they will be contacted via telephone, weekly during first month and fortnightly afterwards to address concerns/issues and also to motivate them to keep compliance at a higher level. At each of these visits, the anthropometry and body composition will be assessed, while blood investigations will be repeated at 6 and 12 months. At each eveluations, one to one meeting will be held.

2.6 Statistics The distribution of metabolic derangements will be described using descriptive statistics. Spearman Correlation Coefficients will be used to assess the relationship between percentage fat and metabolic derangements related to NCD as well as anthropometric measurements and metabolic derangements. Comparisons of mean values of these measurements will be made using t tests.

ELIGIBILITY:
Inclusion Criteria:

* Obese children (based on >+2SD of BMI to age on WHO 2007 standards)

Exclusion Criteria:

* Children not of Sri Lankan origin
* Children who are not planning to live in Sri Lanka during the next one year
* Children with a secondary underlying cause for the overweight/obesity

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 339 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vithanage P Wickramasinghe, MD, PhD, Principal Investigator — University of Colombo
Locations (1):
- Lions Club of Negombo Host, Negombo, Western Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Obese (defined as ≥+2SD of BMI for age, WHO 2007 standards) children of 8-16 years of age were identified through a separate screening programme carried out in all schools in the Negombo educational zone and were invited to participate in this study.
  Study commenced in July 2014
Pre-assignment Details: Selected children were invited to participate in the research and provide clinical service. Consent from parents and assent from children obtained.
  After baseline assessment randomly assigned to receive one of the two management protocols on a 1:1 basis. Children were stratified according to gender and age groups; 8-10.99; 11-16 years
Groups:
- Metformin: 8-10.99 year old children will receive metformin. Initially children will be given 250mg of metformin daily for a week and increased to 250mg twice daily for a week and then to 500 mg twice daily there after. 11-16 year old children will receive 500mg of metformin daily initially for one week which will be increased to 500mg twice daily for a week and then to 1g twice daily. The medication will be continued for 12 months.
  Metformin: A dummy tablet similar to Metformin will be administer to the control group
- Placebo: A placebo tablet which is physically similar to metformin tablets will be given in a similar manner as described above (the placebo is manufactured by the same manufacturer, State Pharmaceutical Manufacturing Corporation)
  Metformin: A dummy tablet similar to Metformin will be administer to the control group
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 166 | 173
Completed | 68 | 82
Not Completed | 98 | 91
Not completed — Lost to Follow-up | 28 | 25
Not completed — Withdrawal by Subject | 64 | 58
Not completed — Stopped on family Practitioner advice | 2 | 5
Not completed — Left the area | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Metformin: 166 were randomized to receive Metformin. After a field survey 500 obese children were identified and invited to this study. 155 declined the invitation so the balance 339 were randomized to receive Metformin (166) and placebo (173).
  Children, 8 to 10.99 years received metformin 250mg daily for a week and increased to 250mg twice daily for a week and thereafter 500 mg twice daily. Eleven to 16 year old children received 500mg of metformin daily for one week and increased to 500mg twice daily for a week and thereafter 1g twice daily. Children were asked to take medication with their morning and evening meals to reduce gastro intestinal side effects and risk of hypoglycaemia
- Placebo: 173 were randomized to receive placebo
  Metformin and placebo were manufactured by the State Pharmaceutical Manufacturing Corporation, Sri Lanka and both tablets look similar except for the active pharmacological compound in one
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 166 | 173 | 339
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.92 (2.3) | 11.95 (2.34) | 11.94 (2.31)
Gender [Count of Participants; unit: Participants]
  Female | 78 | 84 | 162
  Male | 88 | 89 | 177
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.89 (3.53) | 27.57 (3.32) | 27.73 (3.42)
BMI Standard Deviation Score [Median (Standard Deviation); unit: units on a scale] — The BMI SDS is calculated by; (BMI value of the subject - median value of the population)/Standard deviation of the population.
  This will provide how far the measured individuals BMI is deviated from the median in multiples of the SD value of the population. Value could be either positive (if measured value is greater than the median) or a negative value (if measured value is less than the median).
  units on a scale | 2.58 (0.42) | 2.54 (0.42) | 2.56 (0.42)
Percentage fat mass [Mean (Standard Deviation); unit: Percent] | 43.02 (5.14) | 42.88 (5.03) | 42.95 (5.08)
Percentage Fat Mass Standard Deviation Score [Mean (Standard Deviation); unit: units on a scale] — The Percent Fat Mass SDS is calculated by; (Percent FM of the subject - median value of the population)/Standard deviation of the population.
  This will provide how far the measured individuals Percent FM is deviated from the median in multiples of the SD value of the population. Value could be either positive (if measured value is greater than the median) or a negative value (if measured value is less than the median).
  units on a scale | 2.82 (0.42) | 2.81 (0.44) | 2.82 (0.43)

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI and Percentage Fat Mass Standard Deviation Scores After One Year of Treatment With Metformin or Placebo
Description: BMI and Percentage Fat Mass SDS was calculated at baseline and one year after giving Metformin or Placebo. The difference is calculated by subtracting the baseline value from one year value (value at 1 year - value at base line value). Data of the 150 that were followed up throughout the period was included.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: Z score
Groups:
- Metformin: After a field survey 500 obese children were identified and invited to this study. 155 declined the invitation so the balance 339 were randomized to receive Metformin (166)
- Placebo: 173 were randomized to receive placebo
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 68 | 82
Z score
  BMI Z score | -0.370 [-0.44 to -0.303] | -0.22 [-0.284 to -0.159]
  Percentage Fat Mass Z score | -0.139 [-0.207 to -0.070] | -0.065 [-0.130 to -0.005]

2. Secondary Outcome: Change in Fasting Insulin After One Year of Treatment With Metformin or Placebo
Description: Fasting insulin was calculated at baseline and one year after giving Metformin or Placebo. The difference is calculated by subtracting the baseline value from one year value (value at 1 year - value at base line value). Data of the 150 that were followed up throughout the period was included.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: pmol/l
Groups:
- Metformin: After a field survey 500 obese children were identified and invited to this study. 155 declined the invitation so the balance 339 were randomized to receive Metforming (166)
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 68 | 82
pmol/l | -58.08 [-111.68 to -4.55] | -26.48 [-77.3 to 24.37]

3. Secondary Outcome: Change in Insulin Resistance Measured by HOMA-IR After One Year Treatment With Metformin or Placebo
Description: HOMA IR (Homeostatic model -Insulin Resistance) was calculated at baseline and one year after giving Metformin or Placebo. The difference is calculated by subtracting the baseline value from one year value (value at 1 year - value at base line value). Data of the 150 that were followed up throughout the period was included.
  Homeostatic model (HOMA-IR = fasting blood sugar(mmol/l) × fasting insulin(mmol/l) ÷ 22.5)
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 68 | 82
units on a scale | -1.77 [-2.577 to -0.980] | -0.792 [-1.549 to -0.035]

4. Secondary Outcome: Change in Triglyceride Levels After One Year of Treatment With Matformin or Placebo
Description: Triglyceride was measured at baseline and one year after giving Metformin or Placebo. The difference is calculated by subtracting the baseline value from one year value (value at 1 year - value at base line value). Data of the 150 that were followed up throughout the period was included.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: mmol/l
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 68 | 82
mmol/l | -0.33 [-0.45 to -0.22] | -0.14 [-0.25 to -0.04]

5. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Levels After One Year of Treatment With Matformin or Placebo
Description: ALT was measured at baseline and one year after giving Metformin or Placebo. The difference is calculated by subtracting the baseline value from one year value (value at 1 year - value at base line value). Data of the 150 that were followed up throughout the period was included.
Time Frame: One year
Measure: Mean (95% Confidence Interval); unit: Iu/l
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 68 | 82
Iu/l | -0.02 [-0.07 to 0.44] | 0.01 [-0.04 to 0.05]

ADVERSE EVENTS:
Time Frame: 13 months (1 month after stopping treatment)
Groups:
- Metformin: 8-10.99 year old children received metformin. Initially children were given 250mg of metformin daily for a week and increased to 250mg twice daily for a week and then to 500 mg twice daily there after. 11-16 year old children received 500mg of metformin daily initially for one week increased to 500mg twice daily for a week and then to 1g twice daily.
  Children were asked to take medication with their morning and evening meals to reduce gastro intestinal side effects and risk of hypoglycaemia. Effects to medication were evaluated before each dose revision and was monitored for all possible adverse events.
- Placebo: The placebo group was given medication in a similar manner and the number of tablets to be taken each occasion were similar to the treatment group
  Children were asked to take medication with their morning and evening meals to reduce gastro intestinal side effects and risk of hypoglycaemia. Effects to medication were evaluated before each dose revision and was monitored for all possible adverse events.
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/173
Other Adverse Events (participants affected / at risk) | 99/166 | 81/173
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=166) | Placebo (N=173)
Vomiting (Gastrointestinal disorders) | 5 (11) | 8 (8)
Nausea (Gastrointestinal disorders) | 19 (34) | 10 (18)
Anorexia (Gastrointestinal disorders) | 33 (62) | 28 (36)
Diarrhoea (Gastrointestinal disorders) | 16 (18) | 12 (12)
Headache (Nervous system disorders) | 4 (8) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 4 (6) — Non speciifc diffuse pain
Gastro oesophageal reflux like symptoms (Gastrointestinal disorders) | 2 (2) | 2 (2) — Mainly complained of heart burn and epigastric pain
Sleepyness (Nervous system disorders) | 1 (1) | 3 (3) — Its not a true CNS maniestation but probably could be due to low sugar levels or part of headache where children are not clearly express
Vertigo (Nervous system disorders) | 0 (0) | 2 (2) — Probably due to hypoglycaemia state but children many not be able to express clearly them
Faintishness (Nervous system disorders) | 11 (11) | 5 (5) — This could be due to hypoglycaemic symptoms, but children may not be able to distinguish and express vertigo even. Non had fainted
papular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Calf Cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No